CLINICAL TRIAL: NCT00402649
Title: Open-Label Study of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Healthy Children Aged 2 Years to 10 Years
Brief Title: Open-Label Study of H5 Vaccine in Participants of Protocol 04-077
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director, ORA, HHS/NIAID/DMID
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06-0072
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Results first posted 2008-11-24 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2008-05

CONDITIONS: Influenza
Keywords: influenza, A/H5N1, avian influenza, vaccine
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

ARMS (1):
- 1 (Experimental): All subjects will receive at least 2 and up to 3 doses of the vaccine approximately 28 days apart.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)

INTERVENTIONS:
Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur) — Inactivated influenza A/H5N1 vaccine administered via intramuscular (IM) injection; dosage 45-mcg.

SUMMARY:
This study may provide safety information on a flu vaccine given to children and may provide immunogenicity information to add to what was collected in a previous flu vaccine study. Participants will include 55 healthy children, ages 2-10, who participated in 04-077 and received a placebo injection instead of the flu vaccine or were incompletely immunized. The study has 2 purposes: to make sure there are no serious side effects in children and to see how the immune systems react to the vaccine. Study procedures include up to 4 study visits, up to 9 follow-up phone calls, 2 blood samples to be collected during visits 1 and 3, and up to 3 vaccine injections in the arm or thigh muscle. Parents will be given a memory aid card to record side effects, temperatures, and medications. Parents will have the option for the child to receive a 3rd dose of vaccine if offered, at month 6. This booster shot will require a 6-month visit and participation for an additional 6 months.

DETAILED DESCRIPTION:
The recent emergence of novel influenza virus strains in human populations has encouraged efforts to develop vaccines for a potential pandemic. The objectives of this study are to evaluate the safety of intramuscular (IM) subvirion inactivated H5N1 vaccine in healthy children aged 2 through 10 years and to determine the immunogenicity profile of IM subvirion inactivated H5N1 vaccine in healthy children approximately 1 month following receipt of the second of 2 doses of vaccine. Study endpoints include: adverse event (AE) and serious adverse event (SAE) information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessments, as indicated); proportion of subjects achieving a serum hemagglutination inhibition antibody titer of 1:40 against the influenza A/H5N1 virus 28 days after receipt of second dose of vaccine (approximately Day 56); geometric mean titer and the frequency of 4-fold or greater increases in hemagglutination inhibition antibody titers 28 days after receipt of second dose of vaccine (approximately Day 56); and development of serum antibody responses against antigenically drifted variants of influenza H5N1 virus. This study is linked to DMID protocol 06-0072. Up to 55 healthy children, aged 2 through 10 years, who previously participated in DMID 04-077, will be eligible for enrollment in this multimember, open-label, phase I/II clinical trial to receive at least 2 and up to 3 doses of an inactivated influenza A/H5N1 vaccine at a 45-micrograms dose. The vaccine dosage level that will be used in this study was chosen based upon safety and immunogenicity data collected previously in adults and children. The injection volume of the 90-micrograms dose is 1 mL for the vaccine being used in this study, but this is considered unacceptable in this age group. Therefore, the 45-micrograms dose (0.5 ml volume) has been selected. Twenty three subjects who were previously enrolled and assigned to placebo in the DMID 04-077 study (A Randomized, Double-Blinded, Placebo-Controlled, Phase I/II, Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Healthy Children Aged 2 Years Through 9 Years) along with up to 32 subjects from a single site who were incompletely immunized are eligible for enrollment in this study. Vaccine will be administered into the deltoid or (if age appropriate) thigh muscle. All subjects will receive 2 doses of the vaccine approximately 28 days apart. At month 6, subjects' parent(s) or guardian(s) will be called to assess the subjects for serious adverse events. Blood collection for immunogenicity studies will be at the discretion of the parent(s) or legal guardian(s). Should data evaluating a third dose of the influenza A/H5N1 vaccine show enhanced immunogenicity in pediatric subjects participating in DMID 04-077, parents/guardians of subjects who received vaccine will be offered the possibility of a third dose for their participating children.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be male or female, aged 2 through 10 years at enrollment, and must have participated in protocol 04-077 as a placebo recipient or a subject at the UCLA site.
* The subject must be in good health (and not on any chronic medications), as determined by medical history and a history-directed targeted physical examination.
* Parents or guardians of the subject must be able to understand and comply with planned study procedures and be available for all study visits.
* Parents or guardians of the subject must provide written consent prior to initiation of any study procedures, and subject may provide written assent as appropriate.

Exclusion Criteria:

* The subject must not have a known allergy to eggs or other components of the vaccine or sensitivity or allergy to latex.
* The subject must not have a history of asthma or recurrent wheezing.
* The subject must not be undergoing immunosuppression as a result of an underlying illness or treatment.
* The subject must not have an active neoplastic disease or a history of any hematologic malignancy.
* The subject must not be using oral or parenteral steroids, inhaled steroids, or other immunosuppressive or cytotoxic drugs. Note: Subjects on nasal or topical steroids will be allowed to enroll in this study.
* The subject must not have a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* The subject must not receive any other inactivated vaccines within 2 weeks before or after any study vaccine or any other live vaccines within 4 weeks before or after any study vaccine in this study.
* The subject must not have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (these conditions include, but are not limited to, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* The subject must not have a history of severe reactions following immunization with contemporary influenza virus vaccines.
* The subject must not have an acute illness, including an axillary temperature greater than or equal to 100 degrees F or an oral temperature greater than or equal to 101 degrees F within 3 days prior to vaccination.
* The subject must not have received an experimental vaccine or medication within 1 month prior to enrollment in this study, or expect to receive an experimental vaccine, medication, or blood product during the 13-month study period.
* The subject must not have any condition that would, in the opinion of the investigator, place them at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* The subject must not have a history of Guillain-Barré syndrome.
* The subject must not be participating concurrently in another clinical trial aside from DMID 04-077 (either in active phase or in follow-up phase).

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCLA Center For Vaccine Research, Torrance, California
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was offered to the 23 subjects (aged 2-10 years) who were previously enrolled and assigned to placebo at the three clinical sites in the DMID 04-077 study (NCT00133536), along with up to 32 subjects from a single site who were incorrectly dosed in that study.
Groups:
- Inactivated Influenza A/H5N1 Vaccine: All subjects will receive at least 2 and up to 3 doses of the vaccine approximately 28 days apart.
Period: Overall Study
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Started | 35
Completed | 33
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Solicited Adverse Events Among All Subjects
Description: Number of subjects reporting solicited Adverse Events collected on Memory Aid for Days 0-7 post each vaccination for all subjects (systematic assessment), for any and severe severities.
Time Frame: Days 0-7 post each vaccination
Measure: Number; unit: Participants
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Number analyzed (Participants) | 35
Participants
  Elevated Oral Temperature of any severity | 0
  Elevated Oral Temperature - severe | 0
  General Activity of any severity | 10
  General Activity - severe | 1
  Pain of any severity | 19
  Pain - severe | 0
  Mobility of any severity | 5
  Mobility - severe | 0
  Redness of any severity | 4
  Redness - severe | 0
  Swelling of any severity | 4
  Swelling - severe | 0
  Rash of any severity | 0
  Rash - severe | 0

2. Secondary Outcome: Number of Participants With Serum Hemagglutination Inhibition (HAI) Antibody Titers of 1:40 or Greater
Description: Number of subjects achieving serum hemagglutination inhibition antibody titer of 1:40 or greater against the influenza A/H5N1 virus after receipt of two doses of vaccine.
Time Frame: Day 28 after second vaccination
Population: Blood draw was optional - blood collected from 16 participants
Measure: Number; unit: Participants
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Number analyzed (Participants) | 16
Participants | 7

3. Secondary Outcome: Geometric Mean Titer of Hemagglutination Inhibition Antibody Titers
Description: Geometric mean titer of hemagglutination inhibition antibody titers after receipt of two doses of vaccine.
Time Frame: Day 28 after second vaccination
Population: Blood draw was optional - blood collected from 16 participants
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Number analyzed (Participants) | 16
Titer | 20.9 [8.4 to 51.9]

4. Secondary Outcome: Number of Participants With a Four-fold or Greater Increase in Hemagglutination Inhibition Antibody Titers
Description: Number of subjects with a 4-fold or greater increase, relative to baseline, in hemagglutination inhibition antibody titers after receipt of two doses of vaccine.
Time Frame: Day 28 after second vaccination
Population: Blood draw was optional - blood collected from 16 participants post vaccination, but missing baseline assessment for 3 of 16 subjects
Measure: Number; unit: Participants
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Number analyzed (Participants) | 13
Participants | 4

5. Primary Outcome: Occurrence of the Solicited Adverse Event of Body Aches, Solicited Only From Children Age 6-10
Description: Number of subjects reporting solicited Adverse Event of Body Aches, collected on Memory Aid for Days 0-7 post each vaccination for children age 6-10 only (systematic assessment), of any and severe severities.
Time Frame: Days 0-7 post each vaccination
Population: Solicited symptom of Body Aches was collected from subjects age 6-10 only
Measure: Number; unit: Participants
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Number analyzed (Participants) | 26
Participants
  Body Aches of any severity | 6
  Body Aches - severe | 0

6. Primary Outcome: Occurrence of Unsolicited Adverse Events
Description: Number of subjects with spontaneous reports of Adverse Events of any and severe severities. Events reported by more than 5.6% of subjects in any group are reported by MedDRA Preferred Term.
Time Frame: Through Day 28 after second vaccination
Measure: Number; unit: Participants
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Number analyzed (Participants) | 35
Participants
  Vomiting of any severity | 2
  Vomiting - severe | 0
  Gastrointestinal viral of any severity | 2
  Gastrointestinal viral - severe | 0
  Nasopharyngitis of any severity | 2
  Nasopharyngitis - severe | 0
  Upper respiratory tract infection of any severity | 2
  Upper respiratory tract infection - severe | 0
  Headache of any severity | 2
  Headache - severe | 0
  Rhinitis allergic of any severity | 2
  Rhinitis allergic - severe | 0

7. Primary Outcome: Occurrence of Serious Adverse Events
Description: Number of subjects with Serious Adverse Events during the 6 months after the first vaccination.
Time Frame: 6 months after the first vaccination
Measure: Number; unit: Participants
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Number analyzed (Participants) | 35
Participants | 0

ADVERSE EVENTS:
Time Frame: Subjects' parents/guardians recorded solicited symptoms on a memory aid for 8 days (Day 0-7) following each dose. Unsolicited non-serious adverse events were collected for 28 days after each dose and serious adverse events were collected through Day 180.
Description: The solicited symptoms are reported separately after each vaccination. The occurrence of a solicited symptom on any day(s) at any severity within the 8 day period was considered one event.
Arm/Group | Inactivated Influenza A/H5N1 Vaccine
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 26/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Inactivated Influenza A/H5N1 Vaccine (N=35)
Vomiting (Gastrointestinal disorders) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 2 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pain - post dose 1 (General disorders) | 5 (5) — Solicited on the memory aid as "Body aches", limited to subjects aged 6-10 years old
Pain - post dose 2 (General disorders) | 2/32 (2) — Solicited on the memory aid as "Body aches", limited to subjects aged 6-10 years old
Injection site erythema - post dose 1 (General disorders) | 4 (4) — Solicited on the memory aid as "Redness", measured in millimeters
Injection site erythema - post dose 2 (General disorders) | 2/32 (2) — Solicited on the memory aid as "Redness", measured in millimeters
Injection site swelling - post dose 1 (General disorders) | 4 (4) — Solicited on the memory aid as "Swelling", measured in millimeters
Injection site swelling - post dose 2 (General disorders) | 2/32 (2) — Solicited on the memory aid as "Swelling", measured in millimeters
Injection site pain - post dose 1 (General disorders) | 11 (11) — Solicited on the memory aid as "Pain at injection site"
Injection site pain - post dose 2 (General disorders) | 15/32 (15) — Solicited on the memory aid as "Pain at injection site"
Decreased activity - post dose 1 (General disorders) | 6 (6) — Solicited on the memory aid as "General activity level"
Decreased activity - post dose 2 (General disorders) | 5 (5) — Solicited on the memory aid as "General activity level"
Joint range of motion decreased - post dose 1 (Musculoskeletal and connective tissue disorders) | 5 (5) — Solicited on the memory aid as "Mobility of injection site limb"
Joint range of motion decreased - post dose 2 (Musculoskeletal and connective tissue disorders) | 3 (3) — Solicited on the memory aid as "Mobility of injection site limb"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less